CLINICAL TRIAL: NCT02145338
Title: Antibiotic Treatment for Intermittent Bladder Catheterisation: A Randomised Controlled Trial of Once Daily Prophylaxis
Brief Title: Antibiotic Prophylaxis for Clean Intermittent Catheterisation
Acronym: AnTIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: NHS Health Technology Assessment Programme (Other); Newcastle University (Other); Glasgow Caledonian University (Other); University of Aberdeen (Other); Cambridge University Hospitals NHS Foundation Trust (Other); North Bristol NHS Trust (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AnTIC:6672; 2013-002556-32 (EudraCT Number); 11-72-01 (Other Grant/Funding Number: NIHR HTA)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Urinary Tract Infections, Recurrent
Keywords: Urinary tract infection; Clean intermittent self-catheterisation; Antibiotic prophylaxis
MeSH Terms: conditions — Urinary Tract Infections | interventions — Nitrofurantoin; Trimethoprim; Cephalexin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antibiotic prophylaxis (Experimental): Nitrofurantoin or Trimethoprim or Cefalexin. Daily antibiotic prophylaxis: nitrofurantoin 50 mg (or 100 mg dependent on participant weight), or trimethoprim 100 mg, or cefalexin 250 mg.
  Interventions: Drug: Nitrofurantoin or Trimethoprim or Cefalexin
- No prophylaxis (Other): The control arm will be a strategy of no prophylaxis. Participants will self-monitor their symptoms as usual and report to their General Practitioner if they develop symptoms and signs suggestive of UTI requiring treatment.
  Interventions: Other: No prophylaxis

INTERVENTIONS:
Drug: Nitrofurantoin or Trimethoprim or Cefalexin — Antibiotic prophylaxis
  Other Names: Macrodantin
  Arms: Antibiotic prophylaxis
Other: No prophylaxis — Discrete treatment courses of antibiotics as indicated by symptoms or signs of UTI.
  Arms: No prophylaxis

SUMMARY:
This research project is designed to find out whether people who suffer repeated urinary tract infections (UTI) related to the need to empty their bladders intermittently with a fine plastic tube (catheter); a process called clean intermittent self-catheterisation (CISC), benefit from taking continuous daily low-dose antibiotics (antibiotic prophylaxis). The investigators estimate that about 40,000 people in the United Kingdom need to use CISC regularly to empty their bladder either because of nerve damage such as multiple sclerosis or because of failure of the bladder muscle to contract, and of these about 25% (10,000 people) suffer frequent UTI. One way to reduce this problem may be to take a small daily dose of antibiotics and the study aims to find out whether such treatment is effective and worthwhile both for the people who suffer the problem and for the National Health Service (NHS).

The two options to be compared in the trial are firstly, a once daily preventive dose (prophylaxis) of an antibiotic routinely used for this purpose (either nitrofurantoin or trimethoprim or cefalexin), and secondly no prophylaxis. The investigators think that an overall decrease of 20% or more in the frequency of UTI would be large enough for future patients using CISC who get troublesome recurrent UTIs to be offered antibiotic prophylaxis routinely. The investigators will also assess any harm caused by continuous use of antibiotics, particularly side effects for those people taking them and changes in the resistance of bacteria to these antibiotics. The investigators can then work out whether the balance between the benefits and harms make the use of prophylaxis worthwhile to people carrying out CISC and for the NHS as a whole.

DETAILED DESCRIPTION:
The AnTIC trial is a 40-site, pragmatic, patient randomised superiority trial comparing an experimental strategy of once daily antibiotic prophylaxis against a control strategy of no prophylaxis. Both groups will otherwise receive usual care including on demand discrete treatment courses of antibiotic treatment for UTI. The trial will be set in both primary and secondary National Health Service (NHS) care. Participants and their clinicians will not be blinded to the allocated intervention but central trial staff managing and analysing trial data will, as far as possible, be unaware of participant allocation. The investigators will also assess participant perception of benefit firstly by completion of a treatment satisfaction questionnaire on exit and secondly by qualitative analysis of semi-structured interviews on trial completion exploring the views and attitudes of a purposive sample of participants towards the trial intervention. The primary economic analysis will assess the cost per UTI avoided but we will also perform a cost-utility analysis and a contingent valuation study. Bacterial ecological change will be assessed by comparing changes in resistance patterns of E. coli in urine and perianal swabs. The investigators have formulated a recruitment plan to progressively build to a target of 372 participants over 24 months.

The primary objective is to determine the relative clinical effectiveness and cost-effectiveness of an experimental UTI prevention strategy of continuous once-daily prophylactic antibiotic therapy against the control strategy of no prophylaxis in people carrying out intermittent bladder catheterisation who suffer recurrent UTI. Outcomes will be collected over 12 months for each participant and analysed at trial termination according to intention to treat.

Primary objectives are:

* Determine the relative impact on incidence of UTI over 12 months
* Determine the incremental cost per symptomatic UTI avoided

Secondary objectives are:

* Clinical

  * Determine the relative effect on quality of life (QoL) amongst trial participants
  * Measure overall satisfaction with prophylactic antibiotic treatment
  * Assess participants' perception of benefit at 12 months
  * Record adverse effects related to both prophylaxis and treatment antibiotic use
  * Determine relative rates of hospitalisation because of UTI
  * Measure difference in estimated glomerular filtration rate (eGFR) at 12 months
  * Determine rates of asymptomatic bacteriuria at 12 months
  * Assess ecological change in E. coli isolated from urine and perianal swabs
* Economic

  * Measure incremental cost per quality-adjusted life year (QALY) gained through repeated completion of SF-36
  * Assess participants' willingness to pay to avoid a UTI by contingent valuation at end of trial participation and incorporate these data in the economic evaluation using a cost-benefit framework.

The investigators will recruit from the population of adult users of CISC. The setting is NHS hospitals and community sites throughout the UK where CISC use is taught and/or monitored. The investigators expect to randomise at least 372 participants over a 24 month period. For primary outcome purposes, follow up will continue for 12 months after intervention. Participants will be consented separately to submit an additional urine sample and perianal swab six months after trial completion (18-month timepoint) to assess return to baseline of E. coli ecology. Separate consent will also be asked for permission to access clinical records for extended follow up for a further nine years (ten years in total) and for life-long linkage to central NHS databases. Allowing for a four-month analysis phase, the total planned trial duration is 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged ≥ 18 years
* Completed training of CISC and predicted to continue use for at least 12 months
* Able to give informed consent for participation in trial
* Able and willing to adhere to a 12-month follow up period
* Have either suffered at least two episodes of symptomatic UTI related to CISC within last 12 months.
* or at least one episode of UTI requiring hospitalization, or for those previously prescribed prophylactic antibiotic for UTI, have completed a 3-month washout period without antibiotic prophylaxis.
* Able to take a once daily oral dose of at least one of nitrofurantoin, or trimethoprim, or cefalexin
* Intermittent catheterisation may be performed by participant, spouse, or carer
* No restriction on type of catheter used

Exclusion Criteria:

* Age < 18 years
* In learning phase of CISC
* Presence of symptomatic UTI - this will be treated and symptoms resolved prior to randomisation
* Already taking prophylactic antibiotic against UTI and declining 3-month washout period without antibiotic prophylaxis (this will be specifically monitored in the screening log)
* Inability to take any of the three prophylactic antibiotic agents due to multiple drug sensitivities
* Women who intend to become pregnant during planned period of trial participation or who are pregnant or who are breastfeeding
* Previous participation in this study
* Inability to give informed consent or have primary outcome information collected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2017-02-22 (Actual)

PRIMARY OUTCOMES:
Relative incidence of symptomatic antibiotic-treated UTI | 12 months
  Relative incidence of symptomatic antibiotic-treated Urinary Tract Infection between the trial groups over 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pickard, MD, Principal Investigator — Newcastle University
Locations (1):
- Institute of Cellular Medicine, Newcastle University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised study data may be made available on request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: These will be published on the NIHR Journals Library in August 2018
Access Criteria: All data requests should be submitted to the Chief Investigator for consideration. Access to anonymised data may be granted following review.

REFERENCES:
- See also: Trial Website — http://research.ncl.ac.uk/antictrial